CLINICAL TRIAL: NCT04745897
Title: Comparing the Accessibility of the World Health Organization's Tuberculosis Guidelines to the eTB Catalogue of Recommendations: A Two-Arm Superiority Randomized Controlled Trial
Brief Title: Accessibility of the World Health Organization's eTB Catalogue of Recommendations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 7908
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Tuberculosis
Keywords: GRADE; Guidelines; Recommendations; Recommendation Mapping; Evidence Mapping
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eTB Catalogue of Recommendation (eTB) (Experimental): New eTB catalogue of recommendations website (eTB).
  Interventions: Other: eTB Catalogue of Recommendations (eTB)
- World Health Organization Tuberculosis Website (WHO TB) (Active Comparator): Current method of accessing tuberculosis (TB) recommendations using World Health Organization (WHO) website (WHO TB).
  Interventions: Other: World Health Organization Tuberculosis Website (WHO TB)

INTERVENTIONS:
Other: eTB Catalogue of Recommendations (eTB) — eTB Catalogue of Recommendations (eTB)
  Arms: eTB Catalogue of Recommendation (eTB)
Other: World Health Organization Tuberculosis Website (WHO TB) — World Health Organization Tuberculosis Website (WHO TB)
  Arms: World Health Organization Tuberculosis Website (WHO TB)

SUMMARY:
The World Health Organization's Global Tuberculosis Programme (WHO-GTB) issues evidence-informed guideline recommendations on tuberculosis (TB). These recommendations are used by decision-makers, guideline developers and other stakeholders. In an effort to improve the accessibility and usability of these recommendations, a new eTB catalogue of recommendations has been developed. This study aims to compare the accessibility of the new eTB catalogue to the earlier method of accessing recommendations directed through the general WHO website.

DETAILED DESCRIPTION:
This is a two-arm superiority randomized controlled trial. The primary objective is to compare the accessibility of information between the eTB catalogue (intervention) and WHO TB (comparison). Secondary outcomes include understanding of the information, satisfaction of catalogue presentation, and preference toward the catalogue. Current and potential users of TB recommendations will be recruited. Data will be collected using a survey with demographic questions and subsequent 1:1 randomization to the intervention. Superiority will be declared if the mean difference in accessibility is 0.5 or greater for the intervention arm on the seven-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Stakeholders who consider themselves to be users or potential users of tuberculosis (TB) recommendations will be eligible for participation. For the purposes of this trial, a user is defined as someone who has previously accessed TB guidelines, recommendations or policy advice, and a potential user is someone who plans to access TB guidelines, recommendations, or policy advice in the future.
* Participants may be part of any group that has a stake in TB, including the public, healthcare providers, policymakers, or researchers. Participants may be from either low- and middle-income countries (LMIC) or high-income countries (HIC).
* They may also vary in levels of education and previous TB work experience.

Exclusion Criteria:

* Individuals involved in eTB catalogue development.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Accessibility of Information on a Seven-Point Likert Scale | Duration of survey (approximately 10 minutes)
  The primary outcome is the accessibility of information on the eTB catalogue compared to the current WHO TB guidelines. Accessibility is defined as the ability to access and use information. This outcome considers the four following domains: (1) how easy is it to find the information (2) how easy is it to understand the information (3) whether the presentation of this information facilitates decision-making (4) overall accessibility of information. These domains will be measured using a seven-point Likert scale (1 = strongly disagree, 7 = strongly agree). The statements will be: 'It was easy to find the information', 'it was easy to understand the information', 'the information was presented in a way that would help me make a decision', and 'this website was easy to navigate'. The investigators will calculate mean composite values of these four domains for the primary outcome of accessibility, and present the four individual domains as secondary outcomes.

SECONDARY OUTCOMES:
Satisfaction on a Seven-Point Likert Scale | Duration of survey (approximately 10 minutes)
  Satisfaction is defined as a stakeholder's impression of catalogue presentation. This outcome considers the three following domains: (1) home page presentation (2) recommendation list presentation (3) individual recommendation presentation.
  These domains will be measured using a seven-point Likert-scale (1 = very dissatisfied, 2 = dissatisfied, 3 = somewhat dissatisfied, 4 = neutral, 5 = somewhat satisfied, 6 = satisfied, 7 = very satisfied). The questions will be: 'how satisfied are you with presentation of the home page?', and 'how satisfied are you with the presentation of the list of recommendations?', and 'how satisfied are you with the presentation of this individual recommendation?'. The investigators will compare means between the intervention and control groups for each domain.
Understanding with Multiple Choice Questions | Duration of survey (approximately 10 minutes)
  Understanding is defined as the correct comprehension of findings. This outcome will be measured using three multiple-choice questions with four choices and one correct answer. There will be an additional option to select 'not found'. The questions will be: 'what is the recommendation strength?', 'what is the certainty of the evidence?' and 'on which page does the evidence to decision (EtD) table for this recommendation start?'. The proportion of correct responses will be compared between groups.
Preference on a Seven-Point Likert-Scale | Duration of survey (approximately 10 minutes)
  Preference is defined as a greater liking of one platform over the other. Participants will be provided with a demonstration of both platforms. They will subsequently answer the question 'between the WHO Tuberculosis Guidelines (current website), and the eTB Guidelines (alternative website), which do you prefer?'. This response will be measured on a Likert-scale (1 = strongly prefer WHO TB, 2 = prefer WHO TB, 3 = somewhat prefer WHO TB, 4 = same preference for WHO TB and eTB, 5 = somewhat prefer eTB, 6 = prefer eTB, 7 = strongly prefer eTB). The means will be compared between the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Holger J Schunemann, MD, PhD, Study Chair — McMaster University; Micayla N Matthews, BHSc, Principal Investigator — McMaster University; Tamara Lotfi, MD, MPH, Study Director — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matthews M, Lotfi T, Santesso N, Loeb M, Mertz D, Chagla Z, Hajizadeh A, Piggott T, Dietl B, Schunemann HJ. Comparing the usability of the World Health Organization's conventional tuberculosis guidelines to the eTB recommendations map: A two-arm superiority randomised controlled trial. PLOS Glob Public Health. 2022 Oct 14;2(10):e0001166. doi: 10.1371/journal.pgph.0001166. eCollection 2022. PMID 36962671
- See also: eTB Catalogue of Recommendations — https://tuberculosis.evidenceprime.com/